CLINICAL TRIAL: NCT06310798
Title: Outcomes of Inter-organizational Health Planning Between Public Dental Care and Municipal Care Organizations for Older People: A Study Protocol for a Randomized Controlled Study in Sweden
Brief Title: Inter-organizational Health Planning for Older Adults: Public Dental Care and Municipal Care
Acronym: GAPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other); Gothia Forum - Center for Clinical Trial (Other); Chalmers University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dnr. 2020-04603
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Oral Health; Oral Health Related Quality of Life; Participation; Participation, Patient; Health Planning
Keywords: health planning; Oral health; older adults; healthy ageing; patient participation; person-centered care
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: In pairs, DHs within public dental care organization in the West of Sweden will be randomized into test and control groups. Due to geographical concerns, NAs within the same municipal as the test control DHs will be asked to participate. As such, the test-group will consist of 12 DHs and 12 NAs. They will form teams in pairs, and each team will collaborate with 15 older adults each in home settings, who participate in the oral assessments and health planning. The control group will consist of 12 DHs which will perform oral assessments according to dental care remuneration programme - business as usual. It is not mandatory but recommended for NAs to participate in the oral assessments, therefore the number of participating NAs within control group is unknown. In total 360 oral assessments and health planning will be performed within the RCT.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inter-professional team test (Experimental): Dental hygienists, nursing assistants and older adults participating in new model for oral health planning in ordinary home settings.
  Interventions: Behavioral: Inter-professional team test
- Oral health planning control (No Intervention): Dental hygienists, nursing assistants and older adults participating in oral health planning in ordinary home settings (business as usual).

INTERVENTIONS:
Behavioral: Inter-professional team test — Digital Platform Support is used to improve communication and collaboration between the different stakeholders involved in the care of older adults. This platform allows for the sharing of oral health assessments, plans, and recommendations, ensuring all parties have access to the same information and can contribute to the care planning process.
  Person-Centered, Three-Step Model:
  Initial oral health assessments conducted by dental professionals, A person-centered planning process where the needs and preferences of the older adults are prioritized, The implementation of tailored oral health care plans, emphasizing shared decision-making and the active involvement of older adults in their care.
  Educational Component: An important element of the intervention is the provision of a two-day course for nursing and dental staff.
  Arms: Inter-professional team test

SUMMARY:
Patient participation is key for healthy ageing and essential in health planning and decision-making. Oral health is an important but sometimes neglected part of general health and there is little research on health planning in ordinary home settings where older adults, dental and nursing staff participate. It has been concluded that shared tools, such as common documentation, and working in teams enables person-centered care in ordinary home settings. Therefore, this protocol outlines the design of a randomized controlled trial (RCT) measuring and comparing effect of two models of team based oral health planning with a common tool (digital platform) in ordinary home care settings in Sweden. The overall aim of this project is to evaluate a person-centered inter-professional and inter-organizational model for oral health planning supported by a digital platform to enable healthy ageing.

Following ethics approval, a study design was developed guided by the seven action-steps of the knowledge to action framework. In the sixth action-step, older adults within the existing dental care remuneration program in Sweden will serve as a base for the RCT. From there older adults,dental hygienists (DH) and nursing assistants (NA) will be randomized into test and control groups. The test group (n= 12 DH and 12 NA) will participate in a two-day course, where a three-step person-centered oral health model will be taught. Control group will be 12 DH within dental care remuneration program conducting business as usual (with unknown number of NA, due to present guidelines). In total 360 older adults/patients will be asked to participate. Test group and control group will respectively have 180 patients each, as such, each team (DH + NA) have 15 patients. Primary outcomes include diverse oral health aspects - the Revised Oral Assessment Guide and the Geriatric Oral Health Assessment Index. Secondary outcomes include a retrospective record review, a health economic evaluation, Person Centered care Assessment Tool and Oral Hygiene Ability Index. Additionally, qualitative studies from theoretical perspectives of change and learning based on interviews with key stakeholders will be conducted in both test and control group.

DETAILED DESCRIPTION:
The overall aim of this project is to evaluate a person-centered inter-professional and inter-organizational model for oral health planning supported by a digital platform to enable healthy ageing.

The evaluation of the revised team-based model assisted by a digital platform is planned to be conducted as a randomized controlled trial (RCT) .

All participation within the RCT, both in terms of professionals and older adults, will be voluntary and the project will be ethically reviewed. In West Sweden, the public dental care organization (including 3200 dental care professionals) is responsible for performing all oral assessments within the dental care remuneration programme. This guarantees a large empirical base. In pairs, DHs within public dental care organizations in West Sweden will be randomized into test and control groups. Due to geographical concerns, NAs within the same municipality as the test control DHs will be asked to participate. As such, the test group will consist of 12 DHs and 12 NAs. They will form teams in pairs, and each team will collaborate with 15 older adults to conduct oral assessments and health planning in home settings. The control group will consist of 12 DHs where each DH will perform oral assessments according to the dental care remuneration programme - that is, they will conduct business as usual on 15 older adults each. It is not mandatory but recommended for NAs to participate in the oral assessments; therefore, the number of participating NAs within the control group is unknown. In total, 360 oral assessments and health planning sessions will be performed within the RCT.

The test group will participate in a two-day course, where initially an informed consent will be signed by all participates, thereafter they will practise:

* Oral assessments according to Revised oral assessment guide.
* Oral hygiene ability assessments according to Oral Hygiene Ability Index.
* Oral health-related quality of life assessment with the Geriatric Oral Health Assessment Index.
* Shared decision-making according to Ottawa Decision Support Framework.
* Using the digital platform. The course will be both theoretical and practical with elements of reflection. Also, test group management within dental and municipal healthcare will participate in a common half-day course where they will learn about the intervention and the digital platform. A dialogue regarding obstacles and opportunities will facilitate a common understanding and the continued implementation process. They will also set common goals regarding how to support the intervention.

At baseline, two project coordinators (DHs) will collect informed consent from all participants, before the intervention. Thereafter empirical data will be collected. All older adults that participate will be enrolled in the dental care remuneration programme and in home care. Participants within the test and control groups will answer on the following parameters at baseline, which will guide the evaluation.

At baseline:

* Empirical data.
* Mini mental state examination (MMSE-SR).
* Revised oral assessment guide.
* Geriatric Oral Health Assessment Index.

Primary outcomes:

* Older adults' oral health status according to Revised oral assessment guide.
* Older adults self-perception of their oral health-related quality of life according to Geriatric Oral Health Assessment Index.

Secondary outcomes:

* Sure of myself; Understand information; Risk-benefit ratio; Encouragement - test before and after health planning in oral assessments. The Sure of myself; Understanding information; Risk-benefit ration; Encouragement-test is based on four validated questions which describe the older adults' uncertainty about which treatment to choose and aspects contributing to uncertainty about the benefits and risks of each option, what matters most to the older adults, support in making a choice and feeling sure about the best choice.
* Person-Centered care Assessment Tool to measure the professionals' experience of the extent to which the care is experienced as being person-centred.
* All participants' (DHs, NAs and older adults) will be measured by health-related quality of life.
* Oral hygiene ability index, for measuring ability to perform oral hygiene tasks. The oral hygiene ability index should be used when indicated, when Revised oral assessments guide shows 2 or 3 at the variables 'teeth', 'gum', 'saliva' and 'oral mucosa' or if the older adult expresses concerns about difficulties with maintaining oral hygiene.

All scales will be measured in both the test and control groups (relation 1:1). Thereafter, test (n=12) and control (n= 12) groups will conduct 15 oral assessments each in ordinary home settings. The DHs and NAs will individually rate their team performance level after each oral assessment from 1 to 10 (1 = very bad, 10 = excellent). Within the test group, options regarding dental care visits will be i) regular dental care visits, ii) digital consultation, iii) mobile unit at ordinary home settings and iv) doing nothing. Within the control group, the options regarding dental care visits will be 'business as usual', namely, i) regular dental care visits, ii) digital consultation or iii) doing nothing.

Follow-up at 6 months:

* Retrospective records review: Number of records including oral health aspects within municipal care. Number of older adults having established contact with dental care. Number of adults having been scheduled for dental treatment at mobile dental units and what treatment have been conducted.
* The oral health recommendations will be analysed compared to existing evidence-based guidelines and recommendations.
* Older adults' oral health status according to Revised oral assessment guide.
* Older adults' self-perception of oral health according to Geriatric oral health assessment index.
* All participants' (DHs, NAs and older adults) health-related quality of life.

Follow-up at 12 months:

* Oral health status according to Revised oral assessment guide.
* Older adults' self-perception of oral health according to Geriatric oral health assessment index.
* All participants' (DHs, NAs and older adults) health-related quality of life.
* Person-Centered care Assessment Tool. Data analysis Baseline characteristics will be presented as numbers (n). Comparisons between group between baseline and follow-up on primary outcomes (Revised oral assessment guide and Geriatric oral health assessment index) will be presented as means and mean changes, with 95 % confidence intervals (CI). Continuous variables will be analysed by t-test (unpaired for comparison between groups and paired for within group analyses). Comparisons between groups will be analysed using chi-square tests. The pre-chosen level of significance will be p < .05. The oral health risk assessment instrument revised oral assessment guide was used in the power calculation. Revised oral assessment index has a possible score of 2-27. Based on the assumption of a mean difference of 1 (SD 3) between the test and control groups, meaning that test group would improve and that the control group would worsen, the power was calculated to 0.8. According to the power calculation the number of older adults needed was 143 in the test- and control- groups, respectively. Given that the participants are frail older adults, an estimated dropout rate of approximately 25% needs to be taken into account, which means that 180 older adults are needed in the test and control groups respectively. The power-analysis has been conducted with assistance by a statistician (AM).

In parallel, research will be conducted to describe the development of the inter-professional and inter-organizational digital platform. Also, individual interviews are planned with professionals (DHs, NAs and managers), the dental team of the mobile unit (dentist and dental nurse) and older adults within the test and control groups. Further on, a health economic evaluation will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled within the Swedish dental remuneration program and enrolled within municipal care services.

Exclusion Criteria:

* Younger than 65 years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Revised oral assessment guide | Measured at baseline
  Validated instrument for oral health assessments including nine items. Lowest rate: 2 - indicating healthy condition, maximum rate 27 indicating poor oral health.
Revised oral assessment guide | Measured at 6 months after baseline
  Validated instrument for oral health assessments including nine items. Lowest rate: 2 - indicating healthy condition, maximum rate 27 indicating poor oral health.
Revised oral assessment guide | Measured at 12 months after baseline
  Validated instrument for oral health assessments including nine items. Lowest rate: 2 - indicating healthy condition, maximum rate 27 indicating poor oral health.
Geriatric oral health assessment index | Measured at baseline
  Validated instrument for oral health related quality of life including 12 items. Minimum rate 12, maximum rate 60. Higher scores indicate better oral health-related quality of life, while lower scores suggest poorer oral health-related quality of life.
Geriatric oral health assessment index | Measured at 6 months after baseline
  Validated instrument for oral health related quality of life including 12 items. Minimum rate 12, maximum rate 60. Higher scores indicate better oral health-related quality of life, while lower scores suggest poorer oral health-related quality of life.
Geriatric oral health assessment index | Measured at 12 months after baseline
  Validated instrument for oral health related quality of life including 12 items. Minimum rate 12, maximum rate 60. Higher scores indicate better oral health-related quality of life, while lower scores suggest poorer oral health-related quality of life.

SECONDARY OUTCOMES:
Sure of myself; understanding information; risk-benefit ration; encouragement-test | Measured at baseline
  Validated instrument, screening for decisional conflicts during health planning, minimum rate 0; maximum rate 4. Low scores indicate high uncertainty regarding options. High scores indicates no decisional conflict.
Person centered care assessment tool | Measured at baseline
  Validated instrument for assessing person centered care, minimum rate 13; maximum rate 65. Higher total score indicate a higher degree of person-centered care, while lower scores suggest areas for improvement.
Person centered care assessment tool | Measured at 12 months after baseline
  Validated instrument for assessing person centered care, minimum rate 13; maximum rate 65. Higher total score indicate a higher degree of person-centered care, while lower scores suggest areas for improvement.

OTHER OUTCOMES:
Retrospective review of records within municipal health care | Measured at 6 months after baseline
  Number of records including oral health aspects within municipal care. Number of older adults having established contact with dental care. - The oral health recommendations will be analyzed compared to existing evidence-based guidelines and recommendations
Participants experiences of oral health planning in ordinary home settings | Measured 3 months after baseline.
  Individual interviews
Oral hygiene ability index (OHAI) | Measured at baseline
  Validated instrument for oral hygiene ability. The scoring system uses scales from 0 to 4 for each oral hygiene task. Once the individual´s performance on each oral hygiene task is assessed and scored, the total score is calculated by adding up the scores for all tasks. Higher scores generally indicate better oral hygiene ability, while lower scores may suggest limitations or difficulties in performing oral hygiene tasks effectively.
Oral hygiene ability index (OHAI) | Measured at 12 months after baseline
  Validated instrument for oral hygiene ability. The scoring system uses scales from 0 to 4 for each oral hygiene task. Once the individual´s performance on each oral hygiene task is assessed and scored, the total score is calculated by adding up the scores for all tasks. Higher scores generally indicate better oral hygiene ability, while lower scores may suggest limitations or difficulties in performing oral hygiene tasks effectively.
Health related quality of life instrument | Measured at baseline
  Health related quality of life instrument. Scoring involves two steps, participants rate their health status in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, respondents select one level of severity that best describes their health state on the day of the assessment. The levels are from 1 - 5, where 1 = no problems, 5 = Extreme problems. The chosen levels for each dimension are combined to form a health state profile, represented by a five-digit code. For example, a health state profile might be "21114" indicating slight problems in mobility and self-care, moderate problems in usual activities and pain/discomfort, and severe problems in anxiety/depression.
Health related quality of life instrument | Measured at 6 months after baseline
  Health related quality of life instrument. Scoring involves two steps, participants rate their health status in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, respondents select one level of severity that best describes their health state on the day of the assessment. The levels are from 1 - 5, where 1 = no problems, 5 = Extreme problems. The chosen levels for each dimension are combined to form a health state profile, represented by a five-digit code. For example, a health state profile might be "21114" indicating slight problems in mobility and self-care, moderate problems in usual activities and pain/discomfort, and severe problems in anxiety/depression.
Health related quality of life instrument | Measured at 12 months after baseline
  Health related quality of life instrument. Scoring involves two steps, participants rate their health status in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, respondents select one level of severity that best describes their health state on the day of the assessment. The levels are from 1 - 5, where 1 = no problems, 5 = Extreme problems. The chosen levels for each dimension are combined to form a health state profile, represented by a five-digit code. For example, a health state profile might be "21114" indicating slight problems in mobility and self-care, moderate problems in usual activities and pain/discomfort, and severe problems in anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Leonardt, PhD, Principal Investigator — Folktandvården Västra Götaland
Locations (1):
- Folktandvården Västra Götaland, Gothenburg, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data that underlie results in a publication may be shared, if it is possible due to General data protection regulation.
Supporting Information: Study Protocol, ICF
Time Frame: This information will be available in November 2024.
Access Criteria: All researchers within the project will be able to access the data. The study protocol will be submitted to Trials. The informed consent form will be tested at ethical committee.
URL: https://pubmed.ncbi.nlm.nih.gov/16255355/

REFERENCES:
- [Derived] Persson Kylen J, Bjorns S, Hagglin C, Bellander L, Brattback Atzori A, Persson Kylen S, Baar AC, Wijk H. Evaluation of collaborative oral health care planning between older adults and personnel from public dental care and municipal care organizations: a study protocol for a cluster-randomized controlled study in Sweden. Trials. 2025 Feb 18;26(1):57. doi: 10.1186/s13063-025-08753-6. PMID 39966931